CLINICAL TRIAL: NCT06988007
Title: Bone Arches: Performance of Pseudo-scanner Sequences in Segmenting the Extent of the Tumour and in Planning Surgical Resection Using the CT Scan as a Reference
Acronym: SARCOUPE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024/17DEC/563
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-04

CONDITIONS: Sarcoma
Keywords: Imaging; sarcoma; cutting guide; MRI
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Intervention Model Description: Whole body MRI in addition to the classic CT assessment for all participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Whole body MRI (Other): Whole body MRI (ZTE sequence)
  Interventions: Device: Whole body MRI

INTERVENTIONS:
Device: Whole body MRI — Whole body MRI (ZTE sequence)

SUMMARY:
The goal of this exploratory interventional study aims to evaluate the performance of "pseudo-scanner" MRI sequences in delineating the tumor extent within bone sarcomas and its ability to serve as a reference for designing cutting guides and enabling "navigation" during the surgical procedure, thus exploring the possibility of replacing the scanner to minimize exposure to ionizing radiation in patients with sarcoma.

DETAILED DESCRIPTION:
The management of bone sarcomas is complex, and imaging plays an important role in both diagnosis and treatment monitoring. MRI is the method of choice to provide accurate information on the extent of the bone tumor and its relationship to adjacent soft tissues. However, an additional CT scan is routinely performed and combined with MRI images (spatial realignment) using software and relying on manual control and/or correction. This is essential during surgical planning to i) ensure resection with properly defined safety margins and ii) allow for accurate bone reconstruction.ing.

This exploratory interventional study aims to evaluate the performance of "pseudo-scanner" MRI sequences in delineating the tumor extent within bone sarcomas and its ability to serve as a reference for designing cutting guides and enabling "navigation" during the surgical procedure, thus exploring the possibility of replacing the scanner to minimize exposure to ionizing radiation in patients with sarcoma.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of bone sarcoma with surgical indication

Exclusion Criteria:

* Implanted material incompatible with MRI.
* Severe claustrophobia.
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the absolute error of surgical margins | through study completion, an average of year
  The error values observed in the study by Cartiaux et al. to assess the reduction in absolute error of surgical margins obtained when using a computer-assisted cutting procedure (using 3DSide software installed on a laptop belonging to 3Dside, made available to the doctoral student) compared to freehand cutting are used to size the present study. The objective is to compare the absolute error resulting from a cutting procedure assisted by this 3DSide software based on "pseudo-scanner" imaging with that resulting from the same procedure based on standard scanner imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Lecouvet, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (2):
- Belgium (2):
  - Cliniques Universitaires Saint Luc, Brussels
  - Cliniques universitaires Saint-Luc, Brussels

IPD SHARING:
Plan to Share IPD: No
Ethic reason

REFERENCES:
- [Background] Evrard R, Schubert T, Paul L, Docquier PL. Quality of resection margin with patient specific instrument for bone tumor resection. J Bone Oncol. 2022 May 13;34:100434. doi: 10.1016/j.jbo.2022.100434. eCollection 2022 Jun. PMID 35601663
- [Background] Bellanova L, Schubert T, Cartiaux O, Lecouvet F, Galant C, Banse X, Docquier PL. MRI-Based Assessment of Safe Margins in Tumor Surgery. Sarcoma. 2014;2014:686790. doi: 10.1155/2014/686790. Epub 2014 Feb 20. PMID 24701131
- [Background] Cobben DC, de Boer HC, Tijssen RH, Rutten EG, van Vulpen M, Peerlings J, Troost EG, Hoffmann AL, van Lier AL. Emerging Role of MRI for Radiation Treatment Planning in Lung Cancer. Technol Cancer Res Treat. 2016 Dec;15(6):NP47-NP60. doi: 10.1177/1533034615615249. Epub 2015 Nov 19. PMID 26589726
- [Background] Sousa JM, Appel L, Engstrom M, Papadimitriou S, Nyholm D, Larsson EM, Ahlstrom H, Lubberink M. Evaluation of zero-echo-time attenuation correction for integrated PET/MR brain imaging-comparison to head atlas and 68Ge-transmission-based attenuation correction. EJNMMI Phys. 2018 Oct 22;5(1):20. doi: 10.1186/s40658-018-0220-0. PMID 30345471
- [Background] Wiesinger F, Bylund M, Yang J, Kaushik S, Shanbhag D, Ahn S, Jonsson JH, Lundman JA, Hope T, Nyholm T, Larson P, Cozzini C. Zero TE-based pseudo-CT image conversion in the head and its application in PET/MR attenuation correction and MR-guided radiation therapy planning. Magn Reson Med. 2018 Oct;80(4):1440-1451. doi: 10.1002/mrm.27134. Epub 2018 Feb 18. PMID 29457287
- [Background] Lecouvet FE, Vande Berg BC, Malghem J, Maldague BE. Magnetic resonance and computed tomography imaging in multiple myeloma. Semin Musculoskelet Radiol. 2001;5(1):43-55. doi: 10.1055/s-2001-12920. PMID 11371335
- [Background] Lecouvet FE, Boyadzhiev D, Collette L, Berckmans M, Michoux N, Triqueneaux P, Pasoglou V, Jamar F, Vekemans MC. MRI versus 18F-FDG-PET/CT for detecting bone marrow involvement in multiple myeloma: diagnostic performance and clinical relevance. Eur Radiol. 2020 Apr;30(4):1927-1937. doi: 10.1007/s00330-019-06469-1. Epub 2019 Dec 16. PMID 31844960